#### University of Pennsylvania Institutional Review Board 3600 Civic Center Blvd., 9th Floor Philadelphia, PA 19104 Ph: 215-573-2540

(Federalwide Assurance # 00004028)

16-Sep-2025

Janos L Tanyi

Janos.Tanyi@uphs.upenn.edu

Attn:

Elkins, Katie L

Katie.Elkins@pennmedicine.upenn.edu

PRINCIPAL INVESTIGATOR : Janos L Tanyi

TITLE : Single Dose Investigator Initiated Pilot Study to Investigate CYTALUX

(pafolacianine) for Intraoperative Imaging of Patients with Endometrial Cancer

Planned for Surgery

SPONSORING AGENCY : ON TARGET LABORATORIES

PROTOCOL # :859066 REVIEW BOARD :IRB #02

Dear Dr. Janos Tanyi:

IRB approval has been given to the above referenced protocol as of 12-Sep-2025. This study will be due for continuing review on or before 20-Aug-2026.

## Approval by the IRB does not necessarily constitute authorization to initiate the conduct of a human subject research study.

Principal investigators are responsible for assuring final approval from other applicable school, department, center or institute review committee(s) or boards has been obtained. If any of these committees require changes to the IRB-approved protocol and informed consent/assent document(s), the changes must be submitted to and approved by the IRB prior to beginning the research study.

If this protocol involves cancer research with human subjects, biospecimens, or data, you may not begin the research until you have obtained approval or proof of exemption from the Cancer Center Clinical Trials Review and Monitoring Committee.

The revisions, in response to review by the convened IRB, were reviewed and approved.

The following documents were included in this review:

The following documents were included in the response:

- -HSERA Response Submission, confirmation code: eedchjgc, submitted on 9/4/2025
- -Response to IRB Stipulations Letter Dated 03-Sep-2025
- -Response to CTSRMC Stipulations Letter Dated 03-Sep-2025
- -Protocol v3.0 Dated 03-Sep-2025
- -Informed Consent/HIPAA Authorization Form Dated 05-Sep-2025, submitted via email

The following documents, submitted under code: eebeaffj, were previously reviewed by the IRB on 8/21/2025 and are now approved:

- -Cover Letter Dated 8 August 2025
- -OCR IND Exempt Determination Letter Dated 03-Jul-2025
- -CYTALUX (pafolacianine) [OTL38] Investigator's Brochure Edition 4.0 Dated 03-Nov-2023
- -Anatomic Pathology Services Form Dated 04-Aug-2025
- -Lab Services Form Dated 04-Aug-2025
- -Letter of Support Dated 04-Aug-2025

- -CTSRMC Disease Discipline Focus Group Form Dated 04-Aug-2025
- -CTSRMC Justification and Prioritization Form Dated 04-Aug-2025
- -CTSRMC In-House Monitoring Plan Dated 04-Aug-2025

When enrolling subjects at a site covered by the University of Pennsylvania's IRB, a copy of the IRB approved informed consent form with the IRB approved from/to stamp must be used unless a waiver of written documentation of consent has been granted.

If you have any questions about the information in this letter, please contact the IRB administrative staff. Contact information is available at our website: http://www.upenn.edu/IRB/directory.

Thank you for your cooperation.

Sincerely,

Candace Digitally signed by Candace Adams Date: 2025.09.16 14:20:03 -04'00'

IRB Administrator

# UNIVERSITY OF PENNSYLVANIA RESEARCH PARTICIPANT INFORMED CONSENT AND HIPAA AUTHORIZATION FORM

**Protocol Title:** Single Dose Investigator Initiated Pilot Study to Investigate

CYTALUX (pafolacianine) for Intraoperative Imaging of Patients with Endometrial Cancer Planned for Surgery

**Principal** Janos Tanyi, M.D., Ph.D. **Investigator:** 3400 Civic Center Blvd

Perelman Center for Advanced Medicine

3rd Floor West 215-662-3318

**Emergency** 24-Hour Emergency Number: 215-662-4000

**Contact:** Ask for the surgical fellow on call

### **Research Study Summary for Potential Participants**

You are being invited to participate in a research study. Your participation is voluntary, and you should only participate if you completely understand what the study requires and what the risks of participation are. You should ask the study team any questions you have related to participating before agreeing to join the study. If you have any questions about your rights as a human research participant at any time before, during or after participation, please contact the Institutional Review Board (IRB) at (215) 898-2614 for assistance.

The research study is being done to assess the safety and ability of an investigational drug called CYTALUX (pafolacianine) and a special camera system for the detection of cancer in patients undergoing surgical resection for endometrial cancer.

If you agree to join the study, you will be asked to complete the following research procedures:

- Informed consent and HIPAA authorization process;
- Confirmation that you are a surgical candidate.
- Blood draw and/or urine sample for lab test for pregnancy if you are able to become pregnant.
- You will be asked to answer questions about your general health, medical history, and cancer diagnosis information.
- Other information collected as part of your routine care and the screening research procedures, includes age, sex, race, and ethnicity.

Your participation will last for approximately 2 months.

The most common risks of participation are flushing, nausea, vomiting, abdominal pain and itching from the infusion of the CYTALUX (pafolacianine).

Please note that there are other factors to consider before agreeing to participate such as additional procedures, use of your personal information, costs, and other possible risks not discussed here. If you are interested in participating, a member of the study team will review the full information with you. You are free to decline or stop participation at any time during or after the initial consenting process.

### Why am I being asked to volunteer?

You are being invited to participate in a research study because you have endometrial cancer and will be undergoing surgery as a part of treatment. During the surgery for your endometrial cancer, the study doctor tries to remove as much of the cancer as possible from your pelvic and abdominal area. In an attempt to remove the cancer, the study doctor may need to remove the ovaries, the uterus (womb) including the cervix (opening of the womb), the fallopian tubes ("tubes") and/or other organs.

CYTALUX is a special diagnostic product (medicine) made from folate (a type of B vitamin) that's linked to a glowing dye. When it's given to a patient, it should attach to cancer cells because they usually have more folate "receptors" than normal cells. During surgery, doctors use a special camera with near-infrared light to see the glow from the dye, which makes the cancer cells light up. This approach helps surgeons spot cancer more clearly, even tiny or hidden spots that might be missed by the naked eye or by touch alone. This could help the doctor see the cancer better during the surgery, which may help her/him take out additional cancer or the cancer more completely.

Your doctor may be an investigator in this research study. You do not have to participate in any research study offered by your doctor. If you choose not to participate, there will be no loss of benefits to which you are otherwise entitled. You may also decide to discuss the study with your family, friends, or family doctor. Being in a research study is different from being a patient. As an investigator, your doctor is interested both in your clinical welfare and in the conduct of this study.

If you decide to participate, you will be asked to sign this form.

## What is the purpose of this research study?

- See if CYTALUX (pafolacianine) helps light up the endometrial cancer when viewed with the special camera system.
- Test the safety of CYTALUX (pafolacianine) to see if you can tolerate it.

CYTALUX (pafolacianine) and the camera system are approved by the FDA for use in adult patients with ovarian cancer and cancerous and non-cancerous lung lesions. CYTALUX (pafolacianine) and the camera system are considered to be investigational (study drug/device) because your doctor is using them for a different cancer type that is not currently FDA approved as part of the drug and device labels.

### How long will I be in the study?

Your involvement in this study will last approximately 2 months.

In this study, you will have your first visit up to about one month before your surgery. You can receive CYTALUX (pafolacianine) on the day of surgery or up to 7 days before your surgery. You will be followed until about 4 weeks after your surgery.

Up to 10 patients with endometrial cancer may take part in this study. All patients will receive the study drug.

#### What am I being asked to do?

Once your doctor and/or a member of the doctor's team has answered all your questions about the study and you have given written permission to take part in this study by signing this form, your medical history (questions about your health) will be reviewed with you before your surgery to ensure you are able to participate in the study. Your tests done, that are the same as those that are done before any major surgery, will be reviewed. There could be additional lab and/or imaging tests if you experience any side effects from the CYTALUX (pafolacianine). Some of the tests could be done again before, during, and/or after your surgery.

Your participation in this study is divided into different visit types where examinations, tests and your surgery will be performed.

It is important to tell your doctor if you are taking vitamins that contain Folic Acid (vitamin B9), or Folic Acid (vitamin B9) supplements. You will need to stop taking these vitamins at least 48 hours before your scheduled infusion. Folic acid can reduce the effectiveness of the CYTALUX (pafolacianine). Certain other medications have not been studied together with CYTALUX (pafolacianine), so it is important to tell your doctor about all medicines and supplements you are taking.

**Screening Visit** (To see if you can take part in the study and will take place no more than 30 days before your surgery)

During the Screening Visit, the doctor and/or a member of the doctor's team will ask you about your health, and obtain a list of all medications, including vitamins and over-the-counter medications (medicines obtained without a doctor's prescription), that you are taking.

#### **Study Drug Infusion** (Up to 7 days before surgery)

- You will be scheduled to receive the drug being tested, CYTALUX (pafolacianine), any time from 7 days before your surgery up to the day of your surgery. You will receive CYTALUX (pafolacianine) at least one hour before the imaging portion of your surgery.
- Before you receive the study drug, the following will happen:
  - The doctor and/or a member of the doctor's team will ask you about your health and obtain a list of all medications including vitamins and over-thecounter (medicines obtained without a doctor's prescription) medicines that you are taking.
  - For patients who are able to have children, a urine pregnancy test will be done.

 The study drug will be given to you over about 60 minutes through a vein. The dose of CYTALUX (pafolacianine) given to you will be calculated by your weight.

#### **Surgery Visit**

The following activities related to the study will happen on the day of your surgery:

- The doctor will look for cancer as they usually do by feeling and looking throughout your peritoneal cavity using white light and will record the findings.
- After this, the doctor will use the special camera system to look for cancer
  that may light up where the CYTALUX (pafolacianine) has attached and will
  record the findings. Any cancer that is seen with the use of the special
  camera system may be the same as what the doctor recorded earlier without
  the use of the camera system, or there may be additional cancer seen.
- The doctor will then remove the cancer that has been detected, and any areas that they think should be taken out. This removal of the cancer will be done as the doctor would usually do in surgery for endometrial cancer.
- After the doctor has removed the cancer as discussed above, she/he will
  once again use the camera system to see if there is any cancer left and the
  findings will be recorded. Any such cancer observed will be removed based
  on the doctor's judgment.
- The cancer tissue that is removed will be sent to the lab for further testing.
- Any side effects that you may have with the use of CYTALUX (pafolacianine) and/or the camera system will be recorded.
- A sample of any cancer that is removed during this study will be sent to the hospital's laboratory for testing to see if it is endometrial cancer, and to see if the cancer has certain receptors on the surface that would cause the drug, CYTALUX (pafolacianine), to attach to the cancer.

#### Post-operation Visit (Day 28 ± 7 Days)

- About 4 weeks after the surgery, you will be contacted via phone by the doctor and/or a member of the doctor's team, or asked to come to the clinic.
- You will be asked about how you are feeling and about all the medications, including vitamins and over-the-counter (medicines obtained without a doctor's prescription) medicines, that you are taking. The findings will be recorded.

### What are the possible risks or discomforts?

Taking part in this study involves some risks and possible discomfort.

#### Risks of CYTALUX (pafolacianine) and Camera System

The following adverse reactions were reported in patients receiving CYTALUX (pafolacianine) in clinical studies:

- nausea
- vomiting
- abdominal pain
- flushing (redness on face)
- hypersensitivity (very sensitive)
- elevation in blood pressure
- upset stomach
- chest discomfort

A total of 17% (69 out of 406) of patients experienced reactions during administration of Pafolacianine.

Some of the side effects could be due to an allergy-like reaction.

Although not seen in the study of CYTALUX (pafolacianine) in healthy individuals, allergy-like reactions can rarely be severe, and could be serious and life-threatening. Some of the side effects of a severe, serious allergy-like reaction include having the following:

- difficulty breathing
- wheezing
- a sudden drop in blood pressure (making you feel dizzy or lightheaded or feel as if you are passing out)
- swelling around the mouth, throat, or eyes.

Some of the side effects could go away by temporarily stopping the CYTALUX (pafolacianine) infusion and/or by giving medicines commonly used to treat allergies.

Medicines and equipment to treat side effects will be readily available and your study doctor and/or a member of the study doctor's team will treat side effects based on your condition and their clinical judgment.

Study participants with a known allergy to CYTALUX (pafolacianine) will be given medication(s) approximately 30 minutes prior to the start of the infusion. The medication(s) help prevent an allergy-like reaction.

There are potential risks associated with the use of the camera system. There could be injury to the skin or tissue due to any heat produced by the system.

Errors may occur with the use of CYTALUX (pafolacianine) during real-time tumor imaging during surgery to aid in the detection of cancer, including false positives. A false positive is considered an area that may glow when your doctor is imaging to identify additional areas for cancer that may not be cancer. Your doctor will use his best judgement to determine if this is highlighting an area of concern for cancer. Tissue that does not glow in the surgical field does not rule out the presence of cancer. Additionally, glowing may be seen in normal tissues including bowel, kidneys, lymph nodes, and lungs as well as in inflamed tissues when using CYTALUX (pafolacianine).

In a study with patients who had ovarian cancer it was determined that in 20.2% of patients there were small areas that were removed as part of their surgery that were not cancer (false positive). This did not change the safety for these patients who received CYTALUX (pafolacianine).

It is impossible to predict all the possible side effects that may be seen with CYTALUX (pafolacianine) and/or the use of the camera system. As with any drug, unknown risks and side effects are also possible, and you could experience a side effect that has not been anticipated with CYTALUX (pafolacianine) and/or the camera system.

#### Risks of Surgery and Anesthesia (Standard/Usual Care Risks)

The risks and complications associated with the surgery and anesthesia will be reviewed by your physician and outlined in a separate consent form.

Although complications from venipuncture (blood drawing), subcutaneous and intravenous injections occur very rarely, all, some, or none of the following may occur: a bruise or lump at the puncture site, local bleeding, local infection and lightheadedness.

There may be other complications or risks that we do not know about right now.

## Risks associated with delivery of the CYTALUX (pafolacianine) (Study Participation Risks)

You will receive CYTALUX (pafolacianine) directly into a vein through a needle. This may cause the following problems:

- irritation of the vein; you could feel warmth, swelling, pain, or redness around the area near the vein.
- damage to your vein
- damage to the skin or tissue around the injection site
- a blood clot or an air bubble could form, which could block a blood vessel in another part of your body
- infection at the site where the needle is inserted into the vein
- delay of surgery as a result of a reaction to the drug.

## Risks associated with increasing the scale of the operation (Study Participation Risks)

If the surgeon increases the scale of the operation, you may have to stay in the hospital longer than expected or have additional post-operative complications. This can increase the risk of certain infection acquired from extended hospital stays. However, the scale of the operation will not become larger than what you have consented for as a part of your normal clinical care.

The video images that are being taken as part of a research study come with additional risks:

There is a chance that while removing additional tissue that glows in the video images, you could be put at an increased risk of having a surgical complication.

A surgical complication includes, but is not limited to:

Bleeding, infection, pain, injury to a major organ, nerve damage, blood clot in the arms/legs/other region of the body, and death.

There is a chance that being under anesthesia for the additional ten (10) minutes could put you at an increased risk of having a common side effect associated with anesthesia. These common side effects include, but are not limited to:

Nausea and vomiting after surgery, sore throat and hoarseness, shivering/chills, confusion, and muscle aches.

Finally, there is a chance that the imaging technique of the cameras may falsely reassure the surgeon that all of the tumor has been taken out, so not as much tissue will be removed. In other words, not all of the abnormal tissue could be taken out.

Your surgeon will do everything possible to minimize these risks. If your surgeon thinks that removing additional tissue is too risky, they will not remove the additional tissue. Again, there will be no plan of stopping your surgical procedure if the images indicated a possible, distant metastatic disease as this is an experimental procedure.

#### Risks that are not known and risk of pregnancy:

As with any drug, unknown risks and side effects are also possible, and you could experience a side effect that has not been anticipated with the drug, CYTALUX (pafolacianine), being studied in the clinical trial and/or the camera system. There is also a chance that other medications you may be taking could react with CYTALUX (pafolacianine).

For your safety, you must tell the study doctor and/or a member of the doctor's team about all medications you are taking before you start the study and/or during the study. This should include vitamins, nutritional supplements, and over-the-counter medicines (medicines obtained without a doctor's prescription) that you are taking.

#### Reproductive risks

There is not enough information to know what the risks might be to a breast-fed infant or to an unborn child carried by a woman who takes part in this study.

Patients who could become pregnant must agree to use a medically acceptable form of birth control from the time of signing of this consent document until 30 days after the study completion. However, if you are menopausal (without a menstrual period for 2 consecutive years), have had a hysterectomy, or are over the age of 60 you will not be required to take a pregnancy test. If you suspect you are pregnant, you must tell the study doctor immediately.

If there is the possibility of you breast feeding you should not participate in the study. Before initiating any breast feeding, please discuss it with the study doctor.

Women who can become pregnant will have a pregnancy test before taking part in this study. For the pregnancy test, you will give a urine sample within about 24 hours before you get CYTALUX (pafolacianine). You will be told the results of the pregnancy test. If the pregnancy test is positive, you will not be able to take part in the study.

#### Risks of Genetic Testing

This research includes genetic testing. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.

There can be a risk in knowing genetic information. New health information about inherited traits that might affect you or your blood relatives could be found during a research study. Even though your genes are unique, you share some of the same

genes with your blood relatives. Although we are not able to know all of the risks from taking part in research on inherited traits, we believe that the risks to you and your family are very low, because your samples will be coded.

Very rarely health or genetic information could be misused by employers, insurance companies, and others. For example, it could make it harder for you to get or keep a job or insurance, or life insurance companies may charge a higher rate based on this information. We believe the chance these things will happen is very small, but we cannot make guarantees.

A federal law (Genetic Information Non-Discrimination Act, GINA) helps reduce the risk from health insurance or employment discrimination. The law does not include other types of misuse by life insurance or long term care insurance. If you want to learn more about GINA, you can find information about it on the internet or ask the study staff.

#### What if new information becomes available about the study?

During the course of this study, we may find more information that could be important to you. This includes information that, once learned, might cause you to change your mind about being in the study. We will notify you as soon as possible if such information becomes available.

### What are the possible benefits of the study?

You may not get any benefit from being in this research study.

The use the camera during surgery may make your cancer more visible to the surgeon during your surgery, but any benefits of this are not known at present.

The information obtained from this study may eventually be helpful for the treatment of cancer patients in the future.

## What other choices do I have if I do not participate?

You do not have to be in this study to receive treatment, including surgery, for your endometrial cancer. You could undergo the surgery for endometrial cancer without the use of CYTALUX (pafolacianine). You should talk to the study doctor and/or a member of the doctor's team, and/or your regular doctor about each of your choices before you decide if you will take part in this study.

## Will I be paid for being in this study?

You will not be paid for taking part in this study.

### Will I have to pay for anything?

You will not need to pay for tests and procedures (activities) which are done just for this research study. These tests and procedures include:

- CYTALUX (pafolacianine) and giving it to you through a vein
- Testing of the cancer tissue removed for the purpose of this study
- Use of camera system

- However, you and/or your health insurance plan will need to pay for all other tests and procedures that you would normally have as part of the medical care for the endometrial cancer. These tests and procedures include: Scans done before surgery to determine the extent of the cancer
- Surgery and anesthesia
- All pre-operative (before surgery) and post-operative (after surgery) care

Before you agree to be in this study, you should contact your health-care payer/insurer to see if your plan will cover the costs required as part of the care provided by your doctor for the endometrial cancer.

If you have questions regarding billing, insurance or reimbursement for participating in this trial, please contact the study doctor and/or a member of the doctor's team.

#### What happens if I am injured from being in the study?

We will offer you the care needed to treat injuries directly resulting from taking part in this research. We may bill your insurance company or other third parties, if appropriate, for the costs of the care you get for the injury, but you may also be responsible for some of them.

There are no plans for the University of Pennsylvania to pay you or give you other compensation for the injury. If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. You do not give up your legal rights by signing this form.

If you think you have been injured as a result of taking part in this research study, tell the person in charge of the research study as soon as possible. The researcher's name and phone number are listed in the consent form.

For more information on clinical trials and insurance coverage, visit the National Cancer Institute's website at <a href="https://www.cancer.gov">https://www.cancer.gov</a> and type "paying for clinical trials" into the website's search bar. Another way to get this information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

### When is the Study over? Can I leave the Study before it ends?

This study is expected to end after all participants have completed the screening visit, the study drug infusion visit, the day of surgery visit, and the visit 28 days after surgery, and all information has been collected.

This study may also be stopped at any time by your physician, the University of Pennsylvania, or the Food and Drug Administration (FDA) without your consent because:

- The Primary Investigator feels it is necessary for your health or safety. Such an
  action would not require your consent, but you will be informed if such a decision
  is made and the reason for this decision.
- You have not followed study instructions.
- The University of Pennsylvania or the study Principal Investigator, has decided to stop the study.

If you decide to participate, you are free to leave the study at any time. You may do this by contacting the investigator noted on page one of this form. Withdrawal will not interfere with your future care.

#### How will my personal information be protected during the study?

We will do our best to make sure that the personal information obtained during the course of this research study will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. If this study is being overseen by the Food and Drug Administration (FDA), they may review your research records.

If you choose to be in this study, the study doctor will get personal information about you. This may include information that might identify you. The study doctor may also get information about your health including:

- · Past and present medical records
- Research records and results of this clinical study
- Records about phone calls made as part of this research
- Records about your study visits

Information obtained during this research includes medical history and examinations, lab and other test results. Once enrolled in the study, you will be assigned a unique identification number and all your information obtained during this research will identify you by this unique code assigned to you. Only the study investigator and the key research personnel have access to this code list which will be stored on UPHS secured servers and in secure locations accessible to key research personnel only.

Information about your health may be used and given to others, as explained below, by the study doctor and staff. They might see the research information during and after the study.

Information about you and your health, which might identify you, may be given to:

- The U.S. Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- Governmental agencies in other countries
- University of Pennsylvania
- University of Pennsylvania Institutional Review Board (IRB)
- On Target Laboratories, the maker and supplier of CYTALUX (pafolacianine)

Information about you and your health that might identify you may be given to others, as described above, to carry out the research study. The University of Pennsylvania will analyze and evaluate the results of the study.

The information may be given to the FDA. It may also be given to governmental agencies in other countries. The information may also be used to meet the requirements of sending information to governmental agencies.

The results of this research may be published in scientific journals or presented at medical/scientific meetings, but your identity will not be disclosed without your permission.

By signing this consent form, you are giving permission to use and give out the health information listed above for the purposes described above. If you refuse to give permission, you will not be able to be able to participate in this research.

This authorization will not expire unless you withdraw or take away your permission to participate in this research and/or use and disclose your health information at any time. You can do this by sending written notice to the study doctor. If you withdraw your permission, you will not be able to continue being in this study.

When you withdraw your permission, no new health information, which might identify you, will be gathered after that date. Information that has already been gathered may still be used and given to others, as described above. This would be done if it were necessary for the research to be reliable.

Taking part in this research study is voluntary. You can decide not to be in the study and you may decide to stop at any time. You should tell the study doctor and /or a member of the doctor's team if you decide to stop and you will be advised whether any additional tests may need to be done for your safety. In addition, the study doctor may stop you from taking part in this study at any time:

- if the study doctor or study staff believes it is best for you to stop being in the study
- if an unacceptable side effect occurs from the CYTALUX (pafolacianine)
- if you do not follow directions about the study
- if the study is stopped for any reason

If you give permission to give your identifiable health information to a person or business, the information may no longer be protected. There is a risk that your information will be released to others without your permission. Every effort will be made to maintain your confidentiality throughout the study.

### Will information about this study be available to the public?

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## What may happen to my information and samples collected on this study?

#### **Collection of Identifiable Specimens**

Your samples may be used to create products, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

Whole genome sequencing (WGS) will not be conducted on your samples. Whole genome sequencing involves analyzing your entire personal genetic code. WGS can be conducted to determine changes and mutations in DNA. The significance of these results may not be well defined. Not all genetic variations affect one's health.

#### Future Use of Data and/or Specimens

Your information and samples will be de-identified prior to storage for future use. De-identified means that all identifiers have been removed. The information and samples could be stored and shared for future research in this de-identified fashion. The information and samples may be shared with other researchers within Penn, or other research institutions, as well as pharmaceutical, device, or biotechnology companies. It would not be possible for future researchers to identify you as we would not share any identifiable information about you with future researchers. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information and samples only applies to the information and samples collected on this study. If you change your mind, we will not be able to destroy or withdraw your information and samples that were shared because all identifiers would have already been removed.

#### **Electronic Medical Records and Research Results**

#### What is an Electronic Medical Record?

An Electronic Medical Record (EMR) is an electronic version of the record of your medical chart within a health system. An EMR is simply a computerized version of a paper medical record.

If you have never received care within Penn Medicine and are participating in a University of Pennsylvania research study that uses Penn Medicine healthcare related services, an EMR will be created for you for the purpose of maintaining any information produced from your participation. The creation of this EMR is a requirement of your participation in this study. In order to create your EMR, the study team will need to obtain basic information about you that would be similar to the information you would provide the first time you visit a hospital or medical facility (i.e. your name, the name of your primary doctor, the type of insurance you have). If you have been a patient at Penn Medicine in the past, information from your research participation will be added to your existing medical record.

#### What may be placed in the EMR?

Information related to your participation in the research (e.g., laboratory tests, notes from your physician, imaging studies, and clinical procedures, etc.) will be placed in your EMR maintained by Penn Medicine.

Once placed in your EMR your information may be accessible to appropriate Penn Medicine workforce members that are not part of the research team. Information within your EMR may also be shared with others who are determined by Penn Medicine to be appropriate to have access to your EMR (e.g. health insurance company, disability provider, etc).

Penn Medicine also participates in automated information sharing through Health Information Exchanges (HIEs). HIEs securely share parts of your electronic health record, including research information, with other healthcare organizations involved in your care. This information is shared to improve the quality, safety and efficiency of your healthcare. To request that your health information not be shared through HIEs, please call 215-662-4484.

## Will I, as a participant, have access to research related information within the EMR?

The 21st Century Cures Act requires healthcare institutions to allow patients increased access to their electronic medical record. As part of your participation in this research, you will have access to research related information within your EMR through Penn Medicine's patient portal – called MyPennMedicine (MPM).

## Will I receive the results of research testing that may be relevant to my health?

Results that may be relevant to your healthcare will be released to you in your electronic medical record (EMR). These results will be placed in your EMR when the research team receives them.

#### **Incidental Findings**

It is possible that during the course of the research study, the research staff may notice an unexpected finding(s) or information related to your health. Should this occur, the finding(s) will be considered by the appropriate personnel and the PI will inform you if necessary. These possible finding(s) may or may not be significant and may lead to anxiety. You may need to meet with professionals who have the expertise to help you learn more about these results. You can decide whether you want this information to be provided to you. The study team/study will not cover the costs of any follow-up consultations or actions.

## What information about me may be collected, used or shared with others?

The following information may be collected, used or shared with others:

- Name
- Street address, city, county, zip code
- Telephone number
- Medical record numbers
- Health plan ID numbers
- Date of birth
- Demographics such as age, sex, race, etc.
- Personal and family medical history
- Results from physical examinations, tests or procedures

### Why is my information being used?

Your information is used by the research team to contact you during the study. Your information and results of tests and procedures are used to:

- do the research
- oversee the research
- to see if the research was done right
- to evaluate and manage research functions.

### Where may my information be stored?

Information related to your participation in clinical research will be contained in a clinical research management system (CRMS). A clinical research management system (CRMS) is used to register your information as a participant in a study. This allows for your research data to be entered and stored for the purposes of study operational and financial applications and other activities required as part of the conduct of the research. Once placed in the CRMS your information may be accessible to other authorized personnel at Penn Medicine that support research operations. Your information may be held in other research databases.

#### Who may use and share information about me?

The following individuals may use or share your information for this research study:

- The investigator for the study and the study team
- Other authorized personnel at Penn Medicine and the University of Pennsylvania, including offices that support research operations
- Other research personnel with access to the databases for research and/or study coordination and as otherwise approved by the IRB

## Who, outside of Penn Medicine, might receive my information?

#### Oversight organizations

- The U. S. Office of Human Research Protections (OHRP)
- The Food and Drug Administration
- The study data and safety monitoring board

Once your personal health information is disclosed to others outside Penn Medicine, it may no longer be covered by federal privacy protection regulations.

The Principal Investigator or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to Penn Medicine procedures developed to protect your privacy.

## How long may Penn Medicine use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study does not expire.

However, Penn Medicine may not re-use or re-disclose information collected in this study for a purpose other than this study unless:

- You have given written authorization
- The University of Pennsylvania's Institutional Review Board grants permission
- As permitted by law

## Can I change my mind about giving permission for use of my information?

Yes. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the investigator for the study. If you withdraw your permission, you will not be able to stay in this study.

## What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study.

You will be given a copy of this Research Participant HIPAA Authorization describing your confidentiality and privacy rights for this study.

By signing this document, you are permitting Penn Medicine to use and disclose personal health information collected about you for research purposes as described above.

## Who can I call with questions, complaints or if I'm concerned about my rights as a research participant?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research participant, you should speak with the Principal Investigator listed on page one of this form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the IRB at the number on page one of this form.

When you sign this form, you are agreeing to take part in this research study. This means that you have read the consent form, your questions have been answered, and you have decided to volunteer. Your signature also means that you are permitting the University of Pennsylvania to use your personal health information collected about you for research purposes within our institution. You are also allowing the University of Pennsylvania to disclose that personal health information to outside organizations or people involved with the operations of this study.

| _ | Name of Participant (Please Print) Signature of Participant Date | |
|---|---|---|
| _ | Name of Person Obtaining Consent (Please Print) Signature | Date |
| | For participants unable to give authorization, the authorization is gir following authorized participant representative: | ven by |
| | Authorized participant representative Signature | |